CLINICAL TRIAL: NCT06588465
Title: Efficacy of On-venous Laser Irradiation of Blood on Diabetes Kidney Disease Patients: a Single Center, Randomized, Assessor- and Participant-blind, Controlled, Cross-over Clinical Trial
Brief Title: Efficacy of On-venous Laser Irradiation of Blood on Diabetes Kidney Disease Patients
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Yu-Chen Lee, Attending Physician, China Medical University Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: CMUH113-REC1-062
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-05

CONDITIONS: Chronic Kidney Diseases; Proteinuria; Diabetes Mellitus
Keywords: Chronic Kidney Diseases; diabetes mellitus
MeSH Terms: conditions — Renal Insufficiency, Chronic; Proteinuria; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- treatment group A (Experimental): We plan to enroll 72 volunteer patients with microalbuminuria. After 1 week waiting period (as the waiting list group), the patients will be randomized to treatment group A or group B.
  Interventions: Device: On-venous Laser Irradiation of Blood; Device: low dose On-venous Laser Irradiation of Blood
- treatment group B (Experimental): We plan to enroll 72 volunteer patients with microalbuminuria. After 1 week waiting period (as the waiting list group), the patients will be randomized to treatment group A or group B.
  Interventions: Device: On-venous Laser Irradiation of Blood; Device: low dose On-venous Laser Irradiation of Blood

INTERVENTIONS:
Device: On-venous Laser Irradiation of Blood — The treatment will take place three times a week, over six weeks. The On-venous Laser will placed in the body for 60 minutes. A total of 15 laser heads (15 acupoints, bilaterally) will be used in each session.
Device: low dose On-venous Laser Irradiation of Blood — The treatment will take place three times a week, over six weeks. The low dose On-venous Laser will placed in the body for 60 minutes. A total of 15 laser heads (15 acupoints, bilaterally) will be used in each session.

SUMMARY:
The single center, randomized, assessor- and participant-blind, controlled, cross-over on-venous laser irradiation of blood clinical trial was performed to analyze patients with DKD. The information will help to whether integration of laser acupuncture into patient care will help to improve the clinical symptoms and quality of life.

DETAILED DESCRIPTION:
Microalbuminuria is the cardinal symptom of diabetes kidney disease (DKD) and is linked to renal function decline. The cardiovascular risk of patients with DKD is much higher than that of the general population, and cardiovascular diseases is the main cause of death in patients with DKD.

We plan to enroll 72 volunteer patients with microalbuminuria. After 1 week waiting period (as the waiting list group), the patients will be randomized to on-venous laser irradiation of blood and low dose OLIB group. Each group will include 36 patients and given intervention three times a week. The intervention will then be crossed over to the other one after 1 week of wash-our period. Outcome measurement includes questionnaires, biochemistry analysis, urine routine analysis.

ELIGIBILITY:
Inclusion Criteria:

1. HbA1C≥6.5 % and ≤ 9%, ±0.5% under past three months
2. eGFR ≥30ml/min/1.73m2 and protinuria ≥30mg/d under ACEI or ARB treatment

Exclusion Criteria:

1. allergic to laser beans
2. Immunosuppressive drugs had been used in the past six months
3. urine protein over 3.5 g /day
4. Autosomal dominant polycystic kidney disease
5. Lupus nephritis
6. People with mental illness or other mental disabilities are unable to cooperate with the researcher.
7. Those who used non-steroidal analgesics and steroids in the trial period
8. Pregnant or lactating women

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Examine the spot proteinuria changes between the 6th week and at the time of inclusion, as well as between the 13th week and the 6th week. | baseline, 6 weeks, 13weeks
  A spot urine P/C ratio >20 mg/mmol (0.2 mg/mg) is the most commonly reported cutoff value for detecting proteinuria
Examine the eGFR changes between the 6th week and at the time of inclusion, as well as between the 13th week and the 6th week. | baseline, 6 weeks, 13weeks
  eGFR (estimated glomerular filtration rate) is a measure of how well your kidneys are working. Your eGFR is an estimated number based on a blood test and your age, sex, and body type.
Examine the albuminuria changes between the 6th week and at the time of inclusion, as well as between the 13th week and the 6th week. | baseline, 6 weeks, 13weeks
  A ratio of albumin (mcg/L) to creatinine (mg/L) of less than 30 is normal; a ratio of 30-300 signifies microalbuminuria and values above 300 are considered as macroalbuminuria.

SECONDARY OUTCOMES:
SF-36 | baseline, 6 weeks, 13weeks, 17 weeks
  The 36-Item Short Form Survey (SF-36) is outcome measure instrument that is often used, well-researched, self-reported measure of health. It stems from a study called the Medical Outcomes Study for the objective measure of the quality of life.It comprises 36 questions that cover eight domains of health

OTHER OUTCOMES:
The constitution in Chinese medicine questionnaire (CCMQ) | baseline, 6 weeks, 13weeks, 17 weeks
  The CCMQ contain 60 items that consist of the following nine major constitution types: Gentleness (8 Items), Qi- deficiency (8 Items), Yang-deficiency (7 Items), Yin-deficiency (8 Items), Phlegm-damp (8 Items), Damp-heat (6 Items), Blood-stasis (7 Items), Qi-depression (7 Items), and special diathesis (7 Items) types.

CONTACTS AND LOCATIONS:
Overall Officials: YU-CHEN LEE, Ph.D, Study Director — China Medical University, China
Locations (1):
- China Medical University Hospital, Taichung, North Dist, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu S, Zhang F, Bai Y, Huang L, Zhong Y, Li Y. Therapeutic effects of acupuncture therapy for kidney function and common symptoms in patients with chronic kidney disease: a systematic review and meta-analysis. Ren Fail. 2024 Dec;46(1):2301504. doi: 10.1080/0886022X.2023.2301504. Epub 2024 Jan 8. PMID 38189090
- [Background] Chuang SM, Lee CC, Lo WY, Hsieh CL. Effect of acupressure at Sanyinjiao on albuminuria in patients with early diabetic nephropathy: A single-blind, randomized, controlled preliminary study. Explore (NY). 2020 May-Jun;16(3):165-169. doi: 10.1016/j.explore.2019.09.001. Epub 2019 Sep 21. PMID 31591045